CLINICAL TRIAL: NCT06573047
Title: Effect of Thoracic Kineso Tape on Pulmonary Function in Children with Pneumonia
Brief Title: Thoracic KT on Pulmonary Function Ichildren with Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Ali taher elhanfi, Physiotherapist, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: p.t.rec/012/004544
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-08

CONDITIONS: Pneumonia Childhood

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kinesotape (Other): Children in group (b)will receive selected chest physical therapy exercise which including (percussion, huffing, coughing and postural drainage)three times per week for two weeks, each session will be about 20 minutesplus thoracic kinesio-tape every three days (5 times per two weeks). Children will be seated on a chair. When the children will be at the end of the expiration, it will be applied bilaterally on the fifth to sixth and ninth to tenth intercostal muscles transversally and on the anterior and posterior axillary line longitudinally with 50% tension
  Interventions: Other: kinesotape
- chest physiotherapy exercises (Other): the children in the group(a) will receive the selected chest physiotherapy exercise three times per week for two weeks, each session will be about 20 minute which will include the following exercise ( huffing , coughing , percussion,and postural drainage)
  Interventions: Behavioral: Chest physiotherapy exercises

INTERVENTIONS:
Other: kinesotape — a- Kinesio-tape: cure tape (made in Korea) made from 100% gentle cotton fibre and 100% medical grade acrylic adhesive. its Hypoallergenic, water-resistant and does not limit range of motion (ROM), it is come with different colours and sizes. Kinesio Tape is safe enough for a baby's sensitive skin, and gentle enough for aging individuals, flexible enough for rehabilitation, durable enough to support working muscle, joint or ligament and strong enough for athletes at any level.
  Arms: Kinesotape
Behavioral: Chest physiotherapy exercises — selected chest physiotherapy exercise three times per week for two weeks, each session will be about 20 minute which will include the following exercise ( huffing , coughing , percussion,and postural drainage)
  Arms: chest physiotherapy exercises

SUMMARY:
This study aimed to investigate the effect of thoracic kinesio-tape on Pulmonary Functions, time to clinical resolution and respiratory rate and arterial oxygen saturation in children with pneumonia.

Thirty children with pneumonia from both sexes with age ranged from 4 to 7 years participated in this study. The patients were divided into two equal groups (study and control groups), control group received selected chest physiotherapy exercise. Study group received the same selected physical therapy program given to control group in addition to thoracic kinesio-tape three days per week for two weeks.

DETAILED DESCRIPTION:
The study targeted the children with pneumonia (4-7) from both sexes will be selected from tala general hospital in menofia Study design: Randomized controlled trial.

Inclusion Criteria:

1- Children with age between aged 4years to 7 years hospitalized with pneumonia and they assemble all the clinical and radiological criteria for pneumonia 2- Children with stable hemodynamic status 3- Children with no previous history of thoracic surgery, thoracic deformities rib fracture or any condition that make it difficult to apply the KT.

Exclusion criteria:

1. Children with chest drain
2. Children with vision or auditory problems
3. Bone fragility or rib fractures
4. Children with reports of allergic skin reactions to the use of adhesive bandages, plasters, or other adhesive materials
5. Children on ventilator
6. cp children

   I. For Children Selection
   * X-ray to detect the presence of lung infiltrates indicated

   II. For Children Evulation a- Digital spirometer: used to measure pulmonary function include (vital capcity -forced vital capcity -forced expiratory volume1-forced expiratory volume1/forced vital capcity ratio-peak expiratory flow) at the start and at the end of the study.

   B- A pulse oximeter : used to measure oxygen saturation. It is a non-invasive device placed over a person's finger.

   C - The Clinical Respiratory Score (CRS) : The Clinical Respiratory Score appears to have potential as a screening tool for respiratory distress presentations (of several etiologies) in the paediatric emergency department setting of a Low and Middle -Income Countries .Respiratory Score assessed respiratory status in children hospital.

   For treatment

   a- Kinesio-tape made from 100% gentle cotton fibre and 100% medical grade acrylic adhesive. its Hypoallergenic, water-resistant and does not limit range of motion (ROM). Kinesio Tape is safe enough for a baby's sensitive skin, and gentle enough for aging individuals, flexible enough for rehabilitation, durable enough to support working muscle, joint or ligament and strong enough for athletes at any level.

   c- Procedures I. For Children Selection

   - All chest radiographs will be interpreted in the department of radiology (A/P view) and reviewed by pediatric chest physician
   * Children will be clinically evaluated at enrolment of the study and at discharge. A standardized protocol will be taken to record respiratory rate, arterial oxygen saturation.

   II. For Children Evaluation: all children will be evaluated before and after intervention and after 2 weeks from intervention by

1- Pulmonary functions testing: To perform the measurement, subjects will be instructed to sit on an armless chair with back support while their knees flexed to 90° and nostrils will be occluded by a nose clip. Then they will perform a maximal inspiration followed by a forced expiration, exhaling as much air as possible 3 seconds. This maneuver will be repeated 3 times, and the highest scores will be recorded for analyses.

2- Time to clinical resolution which will be defined as the number of days needed for a patient to achieve the following clinical parameters: afebrile (daily maximum body temperature:37.5°C, oxygen saturation :95% and absence of severe signs 3- Respiratory rate and arterial oxygen saturation. A standardized protocol will be taken to record respiratory rate, arterial oxygen saturation. The standard technique for measurement of respiratory rate and arterial oxygen saturation will be the same as previously reported. The daily maximum body temperature was noted by the pediatrician based on the patient's nursing record. The patient's axillary temperature was measured by the attending nurses every 3 hours throughout the hospital stay. All physicians and nurses will be blinded to group assignment and study protocol.

4-The Clinical Respiratory Score (CRS) : The four clinical parameters were : respiratory rate , retractions ,dyspnea and auscultation (table 1) . the score ranged from 1-12 with a higher score indicating more respiratory distress .The score was designed for use while child was awake. the total score obtained there can be 3 categories of respiratory distress: Mild (1- 3), Moderate (4-7), Severe (8-12)

III. Procedures for treatment The control group : the children in the control group will receive the selected chest physiotherapy exercise three times per week for two weeks, each session will be about 20 minutes which included the following exercise;

1. Postural drainage : which involves positioning of the child with the assistance of gravity to mobilize secretions towards the main bronchus .
2. Vibration: In this technique, a rapid vibratory impulse is transmitted through the chest wall from the flattened hands of the therapist by isometric alternate contraction of forearm flexor and extensor muscles, to loosen and dislodge the airway secretions .
3. Percussion: The therapist uses a single hand or both cupped hands or three fingers with the middle finger tented, or a facemask with the port either covered or occluded by a finger, and strikes repeatedly at a rate of three per second over the part of the bronchopulmonary segment that needs to be drained.
4. Huffing: Fast expiration at high volume by the patient .
5. Coughing: Child is requested to cough. In uncooperative or small children, tracheal stimulation or tickling can be performed by placing index finger or thumb on the anterior side of the neck against trachea just above sternal notch with gentle but firm inward pressure in a circular pattern as the child begins to exhale • Thoracic squeezing. This method stimulates the normal cough mechanism through elevation of intrathoracic pressure. This technique, which does not require any special equipment, is used exclusively for the thorax. The hands are placed on the lower third of the thorax. The therapist then applies pressure to increase the forced expiratory volume (FEV) by 30%. It is not necessary to disconnect the patient from the ventilation machine during treatment, which decreases episodes of hypoxemia and the use of high fraction of inspired oxygen (FiO2)

The control Group (B): will receive selected chest physical therapy exercise three times per week for two weeks, each session will be about 20 minutes plus thoracic kinesio-tape every three days (5 times per two weeks). Children will be seated on a chair. When the children will be at the end of the expiration, it will be applied bilaterally on the fifth to sixth and ninth to tenth intercostal muscles transversally and on the anterior and posterior axillary line longitudinally with 50% tension. To stimulate the muscle and support the function, the stimulation technique is usually applied from the origin to the insertion of the muscle with the recommended stretching of 25 to 50%. KT is changed on every third day (for a total of 5 times per two weeks). The children or the care giver will be instructed not to take the tapes off at any time but they will be allowed to take showers. The researcher will complete post treatment evaluations after two weeks for each patient and recorded the data.

ELIGIBILITY:
Inclusion Criteria:

1. Children with age between aged 4 years to 7 years hospitalized with pneumonia and they assemble all the clinical and radiological criteria for pneumonia
2. Children with normal thoracic spine
3. Children with stable hemodynamic status
4. Children with no previous history of thoracic surgery, thoracic deformities rib fracture or any condition that make it difficult to apply the KT.

Exclusion Criteria:

1. Children with chest drain
2. Children with vision or auditory problems
3. Bone fragility or rib fractures
4. Children with reports of allergic skin reactions to the use of adhesive bandages, plasters, or other adhesive materials
5. Children on ventilator
6. cp children

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
pulmonary function | baseline- 5min for each participant
  Vital capacity will carried out by using digital spirometer
Forced vital capacity | baseline- 5min for each participant
  By using digital spirometer
Forced expiratory volume in one second | baseline- 5min for each participant
  By using digital spirometer
Forced vital capacity/forced expiratory volume in one second ratio | baseline- 5min for each participant
  By using digital spirometer
Peak expiratory flow | baseline- 5min for each participant
  By using digital spirometer
Oxygen saturation | baseline- 5min for each participant
  By using oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Sara Elhanfi, Principal Investigator — Cairo University